CLINICAL TRIAL: NCT05075824
Title: A Randomized Double-Blind Phase IIA Study Evaluating the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Crovalimab as Adjunct Treatment in Prevention of Vaso-Occlusive Episodes (VOE) in Sickle Cell Disease (SCD)
Brief Title: A Study Evaluating the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Crovalimab as Adjunct Treatment in Prevention of Vaso-Occlusive Episodes (VOE) in Sickle Cell Disease (SCD)
Acronym: CROSSWALK-c
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BO42451; 2020-004839-25 (EudraCT Number); 2022-502542-28-00 (EU CTIS Number)
Record Dates: First submitted 2021-09-20; First posted 2021-10-13 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Disease
Keywords: Vaso-occlusive episodes; Pain crisis
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Crovalimab (Experimental): Participants will receive a loading series of Crovalimab comprised of an intravenous (IV) loading dose on Day 1, followed by weekly Crovalimab subcutaneous (SC) doses for 4 weeks on Week 1 Day 2, then on Weeks 2, 3 and 4. Maintenance SC dosing will begin at Week 5 and will continue every 4 weeks (Q4W) thereafter for a total of 48 weeks of treatment.
  Interventions: Drug: Crovalimab
- Placebo (Placebo Comparator): Participants will receive matching Placebo administered by IV infusion and SC injection over the same duration as Crovalimab, for a total of 48 weeks of treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Crovalimab — Crovalimab will be administered at a dose of 1000 mg IV (for participants with body weight between 40 kg and 100 kg) or 1500 mg IV (for participants with body weight >= 100 kg) on Week 1 Day 1. On Week 1 Day 2 and on Weeks 2, 3 and 4, crovalimab will be administered at a dose of 340 mg SC. For Week 5 and Q4W thereafter, crovalimab will be administered at a dose of 680 mg SC (for participants with body weight between 40 kg and 100 kg) or 1020 mg SC (for participants with body weight >= 100 kg). Dosing schedule will be as per Arm Description.
  Arms: Crovalimab
Drug: Placebo — Matching Placebo will be administered with the same dosing schedule and equivalent IV and SC volume as weight-based Crovalimab.
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the efficacy, safety and pharmacokinetics of crovalimab compared with placebo as adjunct therapy in the prevention of VOEs in participants with SCD.

ELIGIBILITY:
Inclusion Criteria:

* Body weight >=40 kg.
* Male or female with confirmed diagnosis of HbSS (SCD genotype of sickle cell anemia) or HbSβ0 (SCD genotype of sickle cell beta zero thalassemia).
* Two or more (>=2) to <=10 documented VOEs in the 12 months prior to randomisation.
* If receiving concurrent SCD-directed therapy, the participant must have been on a stable dose for a minimum of 3 months prior to study enrollment. There should be no plans to modify the participants' dosing throughout the study duration, other than for safety reasons.
* If receiving erythropoietin, the participant must have been prescribed this medication for the preceding 3 months and be dose-stabilised for at least 3 months prior to study enrollment.
* Vaccination against N. meningitides serotypes A, C, W, and Y and Vaccinations against H. influenza type B and S. pneumonia.
* Participants who have been vaccinated (partially or in full) against SARS-CoV-2 with a locally approved vaccine are eligible to be enrolled in the study, 3 days or longer after inoculation.
* Adequate hepatic and renal function.
* For women of childbearing potential: agreement to remain abstinent or use contraception during the treatment period and for 10.5 months after the final dose of study treatment.

Exclusion Criteria:

* History of hematopoietic stem cell transplant.
* Participating in a chronic transfusion program and/or planning on undergoing an exchange transfusion during the duration of the study.
* History of hypersensitivity, allergic, or anaphylactic reactions to any ingredient contained in the study treatment.
* Received active treatment on another investigational trial within 28 days (or within five half-lives of that agent, whichever is greater) prior to screening visit, or plans to participate in another investigational drug trial.
* Hemoglobin <6 g/dL.
* Known or suspected hereditary complement deficiency.
* Active systemic bacterial, viral, or fungal infection within 14 days before first drug administration.
* Presence of fever (>=38 degrees Celsius) within 7 days before the first drug administration.
* Immunised with a live attenuated vaccine within 1 month before first drug administration.
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 10.5 months after the final dose of study treatment.
* Known HIV infection with documented CD4 count <200 cells/microliter within 24 weeks prior to screening.
* History of N. meningitidis infection within the prior 6 months.

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2026-04-08 (Estimated)

PRIMARY OUTCOMES:
Annualized rate of medical facility VOEs (AVR) | Baseline up to Week 49

SECONDARY OUTCOMES:
Annualized rate of home VOE | Baseline up to Week 49
Annualized rate of uncomplicated medical facility VOE | Baseline up to Week 49
Annualized rate of Acute Chest Syndrome (ACS) | Baseline to up Week 49
Annualized rate of days hospitalized for medical facility VOE | Baseline up to Week 49
Annualized rate of days hospitalized for treatment of non-VOE complications of SCD | Baseline up to Week 49
Time to first medical facility VOE from randomization | Baseline up to Week 49
Change in urinary albumin-creatinine ratio | Baseline up to Week 49
Change in Tricuspid Regurgitant Jet Velocity (TRV) | Baseline up to Week 49
Percentage of Participants with TRV >2.5 m/s | Week 49
Change in Patient-Reported Outcomes Measurement Information System (PROMIS)-Fatigue Score in Adults | Baseline up to Week 49
Percentage of Participants with Adverse Events (AEs) | Up to 91 weeks
Serum Concentrations of Crovalimab over time | Baseline up to Week 49
Percentage of Participants with Anti-Drug Antibodies to Crovalimab | Baseline up to Week 49

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (27):
- United States (4):
  - Children's Hospital of Michigan, Detroit, Michigan
  - Mississippi Center for Advanced Medicine, Madison, Mississippi
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - East Carolina University, Greenville, North Carolina
- Brazil (8):
  - Hospital Sao Rafael - HSR, Salvador, Estado de Bahia
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - UNESP - Faculdade de Medicina da Universidade Estadual Paulista - Campus Botucatu, Botucatu, São Paulo
  - Hospital das Clínicas Faculdades Médicas de Ribeirão Preto, Ribeirão Preto, São Paulo
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Beneficencia Portuguesa de Sao Paulo, São Paulo, São Paulo
  - HEMORIO, Rio de Janeiro
  - Hospital Samaritano, São Paulo
- CHU Henri Mondor, Créteil, France
- Italy (2):
  - Università degli Studi della Campania Luigi Vanvitelli, Napoli, Campania
  - Azienda Ospedaliera di Verona-Policlinico G.B. Rossi, Verona, Veneto
- Kenya (2):
  - International Cancer Institute (ICI), Eldoret
  - Gertrude's Children Hospital, Nairobi
- Hopital Nini, Tripoli, Lebanon
- Amsterdam UMC Location VUMC, Amsterdam, Netherlands
- Charlotte Maxeke Johannesburg Hospital, Johannesburg, South Africa
- Spain (2):
  - Hospital General Univ. Gregorio Maranon, Madrid
  - Hospital Universitario Miguel Servet, Zaragoza
- Turkey (Türkiye) (3):
  - Adana Acibadem Hospital; Pediatric Hematology, Adana
  - Cukurova University Medical Faculty Balcali Hospital, Adana
  - Mersin Universitesi Tip Fakultesi Hastanesi, Mersin
- United Kingdom (2):
  - Central Middlesex Hospital, London
  - Hammersmith Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing.